CLINICAL TRIAL: NCT06671938
Title: A Phase 2a, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Dosing of Exidavnemab in Patients With Mild to Moderate Parkinson's Disease on Stable Symptomatic Parkinson's Disease Medication and in Patients With Multiple System Atrophy
Brief Title: Safety, Tolerability, and Pharmacokinetics of Exidavnemab in Patients With Parkinson's Disease and Patients With Multiple System Atrophy
Acronym: EXIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BioArctic AB (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAN0805-201; 2024-511222-30-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-19; First posted 2024-11-04 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Parkinson Disease; Multiple System Atrophy
Keywords: Parkinson Disease; Exidavnemab; EXIST; BAN-0805; ABBV-0805; alfa-synuclein
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy

STUDY DESIGN:
Intervention Model Description: The trial will evaluate 2 dose cohorts, dose 1 exidavnemab versus placebo (Cohort 1) and dose 2 exidavnemab versus placebo (Cohort 2). Cohort 2 will consist of a PD cohort (Cohort 2a) and an MSA cohort (Cohort 2b).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants in each cohort will be randomly allocated in a 2:1 ratio to receive either exidavnemab or placebo.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- exidavnemab (Experimental): exidavnemab (cohort 1 - dose 1; cohort 2 - dose 2)
  Interventions: Drug: exidavnemab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Comparator

INTERVENTIONS:
Drug: exidavnemab — The trial medication will be administered as an intravenous (IV) infusion (dose 1; dose 2)
  Arms: exidavnemab
Drug: Placebo Comparator — The trial medication will be administered as an intravenous (IV) infusion
  Arms: Placebo

SUMMARY:
The primary objective of this study is to assess the safety and tolerability of exidavnemab after multiple dosing versus placebo.

DETAILED DESCRIPTION:
This Phase 2a, randomized, double-blind, placebo-controlled, multicenter, multinational, multiple ascending dose (MAD) trial is designed to investigate the safety, tolerability, and pharmacokinetics (PK) of exidavnemab in participants with mild to moderate Parkinson's Disease (PD) on stable symptomatic PD medication and Patients With Multiple System Atrophy.

The trial will evaluate two dose cohorts versus placebo. Participants in each cohort will be randomly allocated in a 2:1 ratio to receive either exidavnemab or placebo. There will be approximately 12 evaluable participants with PD in Cohort 1 and approximately 24 evaluable participants in Cohort 2 (approximately 12 participants in each of Cohorts 2a and 2b), resulting in approximately 36 participants, 24 with PD and 12 with MSA, randomized in total.

ELIGIBILITY:
Inclusion Criteria for Cohorts 1 and 2a (Parkinson's Disease):

1. Male and female participants 40 to 85 years of age.
2. Body weight more than or equal to 50 kg and less than or equal to 120 kg.
3. Have idiopathic PD (i.e., not induced by drugs or other diseases) as defined by bradykinesia combined with at least 1 of resting tremor and rigidity, as per the Movement Disorder Society Criteria for PD (Postuma, et al. 2015).
4. Classified as Stage 1 to 2.5 on the modified Hoehn and Yahr scale for the staging of PD severity.
5. Participants must have cognition inconsistent with dementia as confirmed by a score of more than or equal to 22 on the MoCA.
6. Stable and optimized symptomatic PD medication, defined as the same list of medications for at least 3 months prior to the Screening Visit with no change in the dose for at least 1 month prior to the Baseline Visit, and no planned changes in dose-regimen during trial participation.
7. Prior (any time; i.e., no time limit) or current DaT-SPECT or DaT-PET consistent with dopamine transporter deficit, as per the Movement Disorder Society Criteria for PD(Postuma, et al. 2015). For participants who have not undergone DaT-SPECT or DaT-PET prior to Screening, or who have previously undergone DaT-SPECT or DaT-PET scan(s) but without results consistent with dopamine transporter deficit, DaT-SPECT or DaT-PET should be performed and read locally as part of the Screening procedures.
8. Positive smell test showing hyposmia, as defined by UPSIT scores of around or below the 15% percentile for their relevant sex and age group. Cut-off scores are provided below for reference (Table 5.1; based on Brumm, et al. 2023) Ability to use a tablet device to measure cognitive function, as per Investigator judgment.

Inclusion Criteria for Cohort 2b (Multiple System Atrophy):

1. Male and female participants 40 to 85 years of age.
2. Body weight more than or equal to 50 kg and less than or equal to 120 kg.
3. Have clinically established or clinically probable MSA (either MSA-P or MSA-C), as per the Movement Disorder Society criteria for the diagnosis of MSA (Wenning, et al. 2022).
4. Classified as Stage 1 to 3 on the modified Hoehn and Yahr scale for the staging of MSA severity.
5. Participants must have cognition inconsistent with dementia as confirmed by a score of more than or equal to 22 on the MoCA.
6. Negative urine or serum pregnancy test at the Screening Visit and Baseline for premenopausal women, and for women who have experienced menopause onset less than 12 months prior to the first planned dose of trial medication.
7. Males and POCBP must agree to practice an effective means of birth control during their participation in the trial and until 3 months after their last dose of the trial medication. See specific guidelines regarding contraceptive methods in Section 14.1.
8. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and trial procedures.

Exclusion Criteria for Cohorts 1 and 2a (Parkinson's Disease):

1. Known hypersensitivity to trial medication, the infusion solution, or excipients.
2. More than 5 years of symptomatic treatment for PD.
3. History of neurosurgical intervention for PD including implantation of brain stimulation.
4. Diagnosis of PD dementia or another dementia.
5. Any psychiatric diagnosis or symptoms (e.g., hallucinations, major depression, or delusions) that could interfere with trial procedures.
6. Freezing episodes occurring on a weekly basis or more frequently.
7. Motor fluctuations occurring on a weekly basis or more frequently.
8. Levodopa-induced troublesome dyskinesia of a severity that would significantly interfere with the participant's ability to participate or perform trial procedures as determined by the Movement Disorder Society-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Subscale IV.

Exclusion Criteria for Cohort 2b (Multiple System Atrophy):

1. Known hypersensitivity to the trial medication, the infusion solution, or excipients.
2. Any psychiatric diagnosis or symptoms (e.g., hallucinations, major depression, or delusions) that could interfere with trial procedures.
3. History of significant cardiovascular disease or arrhythmia within 6 months of Screening.
4. Abnormal ECG that is or may be clinically significant in the Investigator's opinion and after consultation with the Medical Monitor, including left bundle branch block, atrial fibrillation, QTcF more than 450 msec for males and more than 470 msec for females at the Screening Visit or Baseline.
5. History of transient ischemic attacks, stroke, or seizures within 12 months of Screening.
6. Abnormal liver function tests: GGT, TBil, ALP, ALT, and AST higher than the ULN and regarded as potentially clinically significant by the Investigator.

   Note: Gilbert's syndrome is not exclusionary.
7. Poorly controlled diabetes as defined by hemoglobin A1C of more than 8%.
8. Contraindication, condition, or concomitant medication incompatible with lumbar puncture (e.g., lumbar scoliosis, coagulopathy, and infected skin at needle puncture site), 1.5T or 3T MRI (e.g., aneurysm clip, metal fragments [e.g., in-skull and cardiac devices other than those approved as safe for use in MRI scanners], and internal electrical devices such as a cochlear implant, spinal cord stimulator, or cardiac pacemaker/defibrillator).

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10-24 (Actual); Primary Completion 2026-03-16 (Estimated); Study Completion 2026-03-16 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events (AEs) and serious adverse events (SAEs). | From first dose to Day 176
  Number of participants with adverse events (AEs) and serious adverse events (SAEs).

SECONDARY OUTCOMES:
Pharmacokinetic (Plasma): Area under the serum concentration-time curve from time zero to the time of the last quantifiable concentration (Clast) | Day 1 and Day 85
  PK parameters (AUClast) following single dose, as calculated by the linear trapezoidal method
Establishment of an appropriate dose range for proof-of-concept trial | From first dose to Day 176
  The recommended maximal dose will be defined by the safety and tolerability profile and PK data
Assessment of systemic immunogenicity effects of exidavnemab | From first dose to Day 176
  Determination of ADAs in serum by using a tier-based approach followed by determination of NAbs if relevant.

CONTACTS AND LOCATIONS:
Locations (8):
- Poland (3):
  - Centrum Medyczyne Neuromed Sp. z o.o., Bydgoszcz
  - Specjalistyczne Gabinety Sp. z o.o., Krakow
  - Krakowska Akademia Neurologii Sp. Z o.o, Krakow
- Spain (5):
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid
  - Policlínica Gipuzkoa, San Sebastián

IPD SHARING:
Plan to Share IPD: No